CLINICAL TRIAL: NCT01855633
Title: Repetitive Transcranial Magnetic Stimulation in Patients With Hemiplegic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dongtan Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Suk Yun Kang, MD, PhD, Dongtan Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-019
Record Dates: First submitted 2013-05-10; First posted 2013-05-16 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tradtional Theta burst stimulation (TBS) rTMS (Experimental): Participants will receive continuous theta burst stimulation (cTBS) rTMS to contralesional hemisphere based on a previous study (Huang et al., 2005)
  Interventions: Device: Traditional Theta burst stimulation (TBS)
- Modified TBS rTMS (Active Comparator): Participants will receive modified cTBS rTMS to contralesional hemisphere based on a previous study (Nyffeler et al., 2006)
  Interventions: Device: Modified TBS rTMS
- Sham rTMS (Sham Comparator): Participants will receive sham cTBS rTMS to contralesional hemisphere.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Traditional Theta burst stimulation (TBS)
  Arms: Tradtional Theta burst stimulation (TBS) rTMS
Device: Modified TBS rTMS
  Arms: Modified TBS rTMS
Device: Sham rTMS
  Arms: Sham rTMS

SUMMARY:
Stroke is one of the major causes of death in the World. Many stroke survivors may suffer from long-term sequelae of stroke such as hemiplegia. The effects of rehabilitation therapy are limited. The development of new treatment strategies is essential. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive method to stimulate the focal area of the brain for restoring brain function. The aim of this study is to investigate the therapeutic effect of rTMS on the motor recovery in patients with hemiplegic stroke.

ELIGIBILITY:
Inclusion Criteria:

* stroke patients with motor weakness
* Medical research council (MRC) grade 0-4
* More than 2 weeks after stroke onset
* Age 18 years and older
* Able to provide consent for the protocol

Exclusion Criteria:

* History of previous symptomatic stroke
* pregnant women
* Persons with surgically or traumatically implanted foreign bodies such as a pacemaker, an implanted medication pump, a metal plate in the skull, or metal inside the skull or eyes (other than dental appliances or fillings), intracardiac lines that may pose a physical hazard during magnetic stimulation will also be excluded
* Patients with history of seizure disorder or epilepsy
* Subjects without the capacity to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-04; Primary Completion 2039-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Keyboard tapping test | 1 day
  Participants will be asked to tap a key of a computer keyboard as fast as possible in five seconds. They will be asked to do three times. We will measure the number of tapping. The primary outcome will be the averaged data of the numbers.This will be done before and after 5-day rTMS intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do, South Korea